CLINICAL TRIAL: NCT06234800
Title: Reasons for Implant Failure and Removal: A Retrospective Study in a Hospital Setting
Brief Title: Observational Study on Implant Removal
Status: Completed | Type: Observational
Sponsor: George Eastman Dental Hospital, Italy (Other)
Responsible Party: Principal Investigator, Lucrezia Paternò Holtzman, Research assistant, George Eastman Dental Hospital, Italy
Other Study IDs: observation study on implant r
Record Dates: First submitted 2024-01-20; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Implant Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Removal of failed dental implants — Removal (with various techniques) of failed dental implants.

SUMMARY:
Reporting of the reason for implant removal in a hospital setting over 20 years. retrospective design.

ELIGIBILITY:
Inclusion Criteria:

* all rehabilitated dental implants

Exclusion Criteria:

* implants with complications that were treated and didn't require removal for complication management.
* patients who could not undergo implant removal for reasons of general health

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients presenting to the department of Oral Surgery with failing or failed osteointegrated dental implants.
Sampling Method: Probability Sample
Enrollment: 381 (Actual)
Dates: Start 2003-01-04 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Implant survival | from 2000 to 2020
  years

CONTACTS AND LOCATIONS:
Locations (1):
- George Eastman Dental Hospital, Roma, Italy

IPD SHARING:
Plan to Share IPD: No
Only means and standard deviations will be shared